CLINICAL TRIAL: NCT02009514
Title: Glucose Control During Glucose Containing And Glucose Free Hemodialysate Evaluated By Continuous Glucose Monitoring In Type 2 Diabetic Patients
Brief Title: Glucose Containing and Glucose Free Hemodialysate in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Pasi I Nevalainen, MD, MD, PhD, Tampere University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R02058M
Record Dates: First submitted 2013-12-03; First posted 2013-12-12 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: End-Stage Kidney Disease; Type 2 Diabetes Mellitus
Keywords: Hemodialysis; Continuous glucose monitoring; Hypoglycemia; Hyperglycemia
MeSH Terms: conditions — Kidney Failure, Chronic; Diabetes Mellitus, Type 2; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Glucose-containing compared to glucose-free hemodialysate — Comparison of effects on glucose variation
  Other Names: Glucose-containing dialysate SK-F 219/1; Glucose-free dialysate SK-F 207

SUMMARY:
The purpose of this study is to investigate differences in glycemia

* during the whole hemodialysis day and the whole freeday
* during hemodialysis, during the evening and the night after hemodialysis and at the same time intervals during the freeday in an unselected type 2 diabetic patient group using both glucose-containing and glucose-free dialysate.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patient
* undergoing stable intermittent thrice weekly hemodialysis for at least one month

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2002-10; Primary Completion 2004-02 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Glucose below 4.0 mmol/l | In the end of a two week period
  In the end of a two-week glucose-containing and glucose-free period percentage of hypoglycemic values of continuous glucose monitoring during the whole hemodialysis day is compared to the whole freeday. Similar comparison is made between the whole glucose-containing and the whole glucose-free hemodialysis day as well as between the whole glucose-containing and the whole glucose-free freeday.

SECONDARY OUTCOMES:
Glucose below 4.0 mmol/l during specified time intervals | In the end of a two-week period
  Percentage of hypoglycemia during the specified time intervals is compared within the glucose-containing and glucose-free hemodialysis day and freeday, and between the glucose-containing and glucose-free hemodialysis day and the freeday. Lastly comparisons are made between the glucose-containing and glucose-free hemodialysis day, and between the glucose-containing and glucose-free freeday.

OTHER OUTCOMES:
Mean glucose | In the end of a two-week period
  Mean glucose of continuous glucose monitoring during the whole glucose-containing and glucose-free hemodialysis day is compared to the whole glucose-containing and glucose-free freeday, respectively. Similar comparison is made between the whole glucose-containing and glucose-free hemodialysis day and between the whole glucose-containing and glucose-free freeday.
Mean glucose during specified time intervals | In the end of a two-week period
  Mean glucose during the specified time intervals is compared within the glucose-containing and glucose-free hemodialysis day and freeday, and between the glucose-containing and glucose-free hemodialysis day and the freeday. Lastly comparisons are made between the glucose-containing and glucose-free hemodialysis day, and between the glucose-containing and glucose-free freeday.
Glucose above 10.0 mmol/l | In the end of a two-week period
  Percentage of hyperglycemic values of continuous glucose monitoring during the whole glucose-containing and glucose-free hemodialysis day is compared to the whole glucose-containing and glucose-free freeday, respectively. Similar comparison is made between the whole glucose-containing and glucose-free hemodialysis day and between the whole glucose-containing and glucose-free freeday.
Glucose above 10.0 mmol/l during specified time intervals | In the end of a two-week period
  Percentage of hyperglycemia during the specified time intervals is compared within the glucose-containing and glucose-free hemodialysis day and freeday, and between the glucose-containing and glucose-free hemodialysis day and the freeday. Lastly comparisons are made between the glucose-containing and glucose-free hemodialysis day, and between the glucose-containing and glucose-free freeday.
Standard deviation of glucose | In the end of a two-week period
  Standard deviation of glucose of continuous glucose monitoring during the whole glucose-containing and glucose-free hemodialysis day is compared to the whole glucose-containing and glucose-free freeday, respectively. Similar comparison is made between the whole glucose-containing and glucose-free hemodialysis day and between the whole glucose-containing and glucose-free freeday.
Standard deviation of glucose during specified time intervals | In the end of a two-week period
  Standard deviation of glucose during the specified time intervals is compared within the glucose-containing and glucose-free hemodialysis day and freeday, and between the glucose-containing and glucose-free hemodialysis day and the freeday. Lastly comparisons are made between the glucose-containing and glucose-free hemodialysis day, and between the glucose-containing and glucose-free freeday.

CONTACTS AND LOCATIONS:
Overall Officials: Pasi I Nevalainen, MD, Principal Investigator — Tampere University Hospital